CLINICAL TRIAL: NCT02424955
Title: Feasibility of 3D Perfusion Ultrasound for Liver Cancer SABR Planning and Response Evaluation
Brief Title: Feasibility 3D Perfusion Ultrasound for Liver Cancer SABR Planning and Response Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-30071; IRB-30071 (Other: Stanford IRB); HEP0048 (Other: OnCore)
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Liver Cancer; Liver Tumor; Hepatocellular Carcinoma; Liver Carcinoma
Keywords: Liver cancer; Hepatocellular Carcinoma; Liver imaging; Stereotactic Ablative Radiotherapy; SABR
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3D Perfusion Ultrasound (Experimental): undergo 3D ultrasound perfusion imaging with perflutren
  Interventions: Drug: perflutren lipid microspheres; Diagnostic Test: 3D ultrasound

INTERVENTIONS:
Drug: perflutren lipid microspheres
  Other Names: Definity
Diagnostic Test: 3D ultrasound

SUMMARY:
The purpose of this study is to prospectively analyze the value of 3D ultrasound perfusion imaging for treatment planning, the prediction of therapy success, and to monitor the treatment response in patients with a primary or metastatic liver tumor undergoing radiation treatment.

DETAILED DESCRIPTION:
Primary Objective:

The primary objectives of this prospective pilot study is to:

1. determine the feasibility and reproducibility of 3D contrast enhanced ultrasound imaging in liver cancer patients undergoing Stereotactic Ablative Radiotherapy and
2. evaluate whether there are treatment induced early changes in imaging metrics derived from 3D contrast enhanced ultrasound. This study will provide valuable insight as to the potential of baseline and/or early post-treatment 3D ultrasound perfusion characteristics (measurements of blood-flow) of primary and metastatic liver tumors to predict tumor response to Stereotactic Ablative Radiotherapy. The investigators' underlying goal is to assess whether early perfusion changes at 1-7 days after SABR initiation can be used as a non-invasive early biomarker for treatment response assessment.

Secondary Objectives:

Evaluate the feasibility of contrast-enhanced ultrasound-to-CT fusion by assisting three-dimensional (3D) perfusion ultrasound (US) imaging with optical and electromagnetic tracking of the ultrasound probe on patients with liver cancer that will undergo CT for treatment planning and/or response evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign the written informed consent document
* Patient with primary liver tumor or metastasis scheduled for Stereotactic Ablative Radiotherapy (SABR)
* Patient is at least 18 years of age. No gender/race-ethnic restrictions.
* Performance status (ECOG) between 0-3
* History and Physical done within 4 weeks of enrollment.

Exclusion Criteria:

* Patient has previously been enrolled in and completed this study.
* Known right to left cardiac shunt, bidirectional or transient.
* Patient has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.
* History of hypersensitivity to the contrast agent perflutren
* History of pulmonary hypertension
* Patients who are pregnant or are trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T. Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3D Perfusion Ultrasound: Patients undergo 3D ultrasound perfusion imaging with perflutren lipid microspheres
Period: Overall Study
Arm/Group | 3D Perfusion Ultrasound
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3D Perfusion Ultrasound
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  50-59 | 3
  60-69 | 2
  70-79 | 5
  80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Perfusion (Blood Volume)
Description: The purpose of this pilot project is to prospectively analyze the value of 3D ultrasound perfusion imaging for treatment planning, the prediction of therapy success, and to monitor the treatment response in patients with a primary or metastatic liver tumor undergoing radiation treatment.
Time Frame: Baseline (pre-treatment), 0-7 days post treatment, 2-4 months post treatment.
Population: No cases were analyzed; analysis was not possible due to poor image quality.
Arm/Group | 3D Perfusion Ultrasound
Number analyzed (Participants) | 0

2. Primary Outcome: Changes in Blood Perfusion (Mean Flow Velocity)
Description: as for outcome 1
Time Frame: Baseline (pre-treatment), 0-7 days post treatment, 2-4 months post treatment.
Population: No cases were analyzed; analysis was not possible due to poor image quality.
Arm/Group | 3D Perfusion Ultrasound
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in Blood Perfusion (Relative Blood Flow)
Description: as for outcome 1
Time Frame: Baseline (pre-treatment), 0-7 days post treatment, 2-4 months post treatment.
Population: No cases were analyzed; analysis was not possible due to poor image quality.
Arm/Group | 3D Perfusion Ultrasound
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | 3D Perfusion Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT02424955/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02424955/ICF_000.pdf